CLINICAL TRIAL: NCT02332096
Title: Screening for Sleep Apnea in Patients Undergoing Atrial Fibrillation Ablation
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Patricia Tung, Instructor in Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2015P000038
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea; Cardiac Arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Atrial Fibrillation: We propose to enroll 100 patients with symptomatic paroxysmal or persistent AF without a known diagnosis of sleep apnea who are referred for an AF ablation procedure at BIDMC. All enrolled subjects will undergo pre-procedure screening sleep study using the Berlin questionnaire and home sleep study using an FDA approved home sleep testing device (HST).
  Interventions: Device: Home Sleep Testing Device

INTERVENTIONS:
Device: Home Sleep Testing Device — Patients will undergo obstructive sleep apnea screening with a FDA approved home sleep testing device.

SUMMARY:
Diagnosis and treatment of sleep apnea with continuous positive airway pressure (CPAP) therapy has been shown to decrease arrhythmia recurrence in patients with AF following ablation. However, patients with AF undergoing ablation are not routinely screened for sleep apnea, despite an estimated sleep apnea prevalence of 25% in the general population, and perhaps higher among patients with AF. Home sleep testing is frequently used for evaluation of sleep apnea.

DETAILED DESCRIPTION:
The American Academy of Sleep Medicine considers atrial fibrillation (AF) to be high risk for sleep disordered breathing, and recommends that those with AF be evaluated for sleep apnea in its clinical guidelines. However, this has not yet become standard practice. The primary reasons for this are that sleep apnea remains under-suspected and under-diagnosed by electrophysiology physicians treating patients with AF, overnight sleep studies are cumbersome and are frequently associated with patient discomfort and high cost, and a mechanism for coordinating sleep apnea screening and treatment referral has not been established in electrophysiology clinics.

The gold standard for the diagnosis of sleep apnea is overnight polysomnography, typically conducted in a sleep laboratory, which can be costly and cumbersome for patients. Home sleep studies are FDA-approved for the diagnosis of sleep apnea and offer patients the opportunity to be assessed in a more natural sleep environment, and often in a more timely manner.

It has been demonstrated that diagnosis and treatment of sleep apnea reduces the risk of arrhythmia recurrence following AF ablation to a level comparable to those without sleep apnea. The goal of this study is to examine the feasibility of screening all patients undergoing AF ablation for sleep apnea, and to refer those patients with sleep apnea for evaluation and treatment by a sleep specialist.

ELIGIBILITY:
Inclusion criteria for the study include:

1. Patients age 18 years and older.
2. Patients with the diagnosis of atrial fibrillation presenting for clinical ablation procedure.

Exclusion criteria for the study include:

1. Patients with an existing diagnosis of sleep apnea.
2. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose to enroll 100 patients with symptomatic paroxysmal or persistent AF without a known diagnosis of sleep apnea who are referred for an AF ablation procedure at BIDMC. All enrolled subjects will undergo pre-procedure screening sleep study using the Berlin questionnaire and home sleep study using an FDA approved home sleep testing device (HST).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-06; Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep apnea in patients with atrial fibrillation | Enrollment

SECONDARY OUTCOMES:
Arrhythmia recurrence | 3 Months
Arrhythmia recurrence | 6 Months
Arrhythmia recurrence | 9 Months
Need for antiarrhythmic medications | 3-12 Months
CPAP compliance when prescribed | 3-12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Tung, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No